CLINICAL TRIAL: NCT05148897
Title: Study of Awareness of Gestational Diabetes Problem Among Sohag Governorate Women
Brief Title: Awareness of Gestational Diabetes Among Sohag Governorate Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Islam Emad Mohamed, Resident doctor at department of internal medicine, Sohag University
Other Study IDs: Soh-Med-21-11-05
Record Dates: First submitted 2021-11-10; First posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Women can participate: among 500 women, over 6 months by random selection and they will be asked to answer the questions of prepared and copied questionnaire sheet.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — a self-administered questionnaire. Based on extensive literature review no questionnaire was found that specifically related to knowledge evaluation. The basic theme of the questionnaire was taken from Diabetes Knowledge Questionnaire (DKN), a well validated tool for knowledge assessment among type 1 and type 2 diabetes mellitus patients. Some modifications were made and new questions particularly related to GDM were included.

SUMMARY:
The type of the study is a cross sectional descriptive using questionnaire method in Sohag governorate among 500 Women, over 6 months by random selection and they will be asked to answer the questions of prepared and copied questionnaire sheet.

Inclusion criteria: all women can participate in this questionnaire.

DETAILED DESCRIPTION:
the study is a cross sectional descriptive using questionnaire method in Sohag governorate among 500 women, over 6 months by random selection and they will be asked to answer the questions of prepared and copied questionnaire sheet. Data was collected by using a self-administered questionnaire. Based on extensive literature review no questionnaire was found that specifically related to knowledge evaluation. The basic theme of the questionnaire was taken from Diabetes Knowledge Questionnaire (DKN), a well validated tool for knowledge assessment among type 1 and type 2 diabetes mellitus patients. Some modifications were made and new questions particularly related to Gestational Diabetes Mellitus (GDM) were included. Final version of questionnaire consists of 15questions divided into five main categories which are basic knowledge about GDM(3 questions), risk factors (3 questions), food and diet values (3 questions), management(3 questions)and complications/outcomes (3 questions). All questions were in multiple choice format with one option was "I don't know "to avoid unnecessary guesses by the participants. Score 1 was given to every right answer and 0 to every wrong answer. A higher score indicates better knowledge about GDM. Thus the maximum score is 15 and minimum is 0 and other questions without score to know the patient himself and to assess the relationship between the residency, work, education level and knowledge of patient and family history.

A standardized questionnaire will focus on:

1. Personal Data
2. Basic Knowledge about GDM
3. Knowledge about risk factors of GDM
4. Knowledge about diet/food values
5. Knowledge about management of GDM
6. Knowledge about GDM complications/outcomes

ELIGIBILITY:
Inclusion Criteria:

* All Females

Exclusion Criteria:

* There is no Exclusion Criteria:

Min Age: 13 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Femalesare the direct face of gestational diabetes, and they are the most vulnerable to the disease and need to be aware of it
Study Population: cross sectional descriptive using questionnaire method in Sohag governorate among 500Women, over 6 months by random selection
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate general knowledge of women about different aspects of Gestational Diabetes: Questionnaire | Change the literacy of knowledge of women about different aspects of Gestational Diabetes at 6 months after the questionnaire
  All the statistical analysis will be done by using Statistical Package for Social Sciences (SPSS Inc., Chicago, IL) version20. Number and percentage will be used for grouped variables whereas mean and standard deviation will be used for continuous variables. Responses to all questions of the questionnaire will be recorded in numbers and percentages. Association of demographic characteristics with knowledge score

CONTACTS AND LOCATIONS:
Overall Officials: Adel A Elsayed, Prof, Study Chair — Professor doctor at department of Internal medicine
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
knowledge of women about different aspects of Gestational Diabetes Mellitus including general knowledge about the disease, risk factors, diet in diabetic patients and complications among the women in Sohag governorate ad the questionnaire itself

REFERENCES:
- [Background] Atlas, D.J.I.D.A., 9th: International Diabetes Federation, International diabetes federation. 2020
- [Background] Eltoony, L.F., et al., Prevalence and Risk Factors for Gestational Diabetes in Aswan, Egypt According to International Association of the Diabetes and Pregnancy Study Groups (IADPSG). 2021. 82(4): p. 701-707.
- [Result] O'Sullivan EP, Avalos G, O'Reilly M, Dennedy MC, Gaffney G, Dunne F; Atlantic DIP collaborators. Atlantic Diabetes in Pregnancy (DIP): the prevalence and outcomes of gestational diabetes mellitus using new diagnostic criteria. Diabetologia. 2011 Jul;54(7):1670-5. doi: 10.1007/s00125-011-2150-4. Epub 2011 Apr 15. PMID 21494772
- [Result] Farrar D. Hyperglycemia in pregnancy: prevalence, impact, and management challenges. Int J Womens Health. 2016 Sep 20;8:519-527. doi: 10.2147/IJWH.S102117. eCollection 2016. PMID 27703397
- [Result] Metzger BE, Coustan DR. Summary and recommendations of the Fourth International Workshop-Conference on Gestational Diabetes Mellitus. The Organizing Committee. Diabetes Care. 1998 Aug;21 Suppl 2:B161-7. No abstract available. PMID 9704245
- [Result] Khan R, Bisnath J, Blackmann J, Bissessar R, Bidhesi S, Boodoo N, Bobb T, Benjamin J, Mohammed A, Mahabir A. Prevalence rates of impaired glucose tolerance and gestational diabetes mellitus amongst expectant mothers and undiagnosed diabetes mellitus in walk-in patients at health centres in North Central Trinidad. J Family Med Prim Care. 2020 Jun 30;9(6):3112-3118. doi: 10.4103/jfmpc.jfmpc_124_20. eCollection 2020 Jun. PMID 32984182
- [Result] Muche AA, Olayemi OO, Gete YK. Prevalence and determinants of gestational diabetes mellitus in Africa based on the updated international diagnostic criteria: a systematic review and meta-analysis. Arch Public Health. 2019 Aug 6;77:36. doi: 10.1186/s13690-019-0362-0. eCollection 2019. PMID 31402976
- [Result] Hegazi R, El-Gamal M, Abdel-Hady N, Hamdy O. Epidemiology of and Risk Factors for Type 2 Diabetes in Egypt. Ann Glob Health. 2015 Nov-Dec;81(6):814-20. doi: 10.1016/j.aogh.2015.12.011. PMID 27108148
- [Result] Cavanaugh KL. Health literacy in diabetes care: explanation, evidence and equipment. Diabetes Manag (Lond). 2011 Mar;1(2):191-199. doi: 10.2217/dmt.11.5. PMID 21860659
- [Result] Lee KW, Ching SM, Ramachandran V, Yee A, Hoo FK, Chia YC, Wan Sulaiman WA, Suppiah S, Mohamed MH, Veettil SK. Prevalence and risk factors of gestational diabetes mellitus in Asia: a systematic review and meta-analysis. BMC Pregnancy Childbirth. 2018 Dec 14;18(1):494. doi: 10.1186/s12884-018-2131-4. PMID 30547769
- [Result] Chu SY, Callaghan WM, Kim SY, Schmid CH, Lau J, England LJ, Dietz PM. Maternal obesity and risk of gestational diabetes mellitus. Diabetes Care. 2007 Aug;30(8):2070-6. doi: 10.2337/dc06-2559a. Epub 2007 Apr 6. PMID 17416786
- [Result] Cheung NW. The management of gestational diabetes. Vasc Health Risk Manag. 2009;5(1):153-64. doi: 10.2147/vhrm.s3405. Epub 2009 Apr 8. PMID 19436673
- [Result] Hussain Z, Yusoff ZM, Sulaiman SA. Evaluation of knowledge regarding gestational diabetes mellitus and its association with glycaemic level: A Malaysian study. Prim Care Diabetes. 2015 Jun;9(3):184-90. doi: 10.1016/j.pcd.2014.07.007. Epub 2014 Aug 15. PMID 25132140